CLINICAL TRIAL: NCT00711139
Title: Phase Ib Follow-up Study to Evaluate Long-term Safety and Tolerability of Immunization With AFFITOPE AD01 Applied During AFFiRiS 001
Brief Title: Long-term Safety and Tolerability of AFFITOPE AD01
Status: Completed | Type: Observational
Sponsor: Affiris AG (Industry)
Responsible Party: Affiris AG
Other Study IDs: Affiris 003; EudraCT 2008-001455-22
Record Dates: First submitted 2008-07-04; First posted 2008-07-08 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer; Morbus Alzheimer; Alzheimer Vaccine; Vaccine; AD; A-beta immunotherapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: AFFITOPE AD01
- 2: AFFITOPE AD01 + Adjuvant

SUMMARY:
The purpose of this study is to assess the long-term tolerability and -safety of AFFITOPE AD01 applied during AFFiRiS 001

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by the patient or the patient's legal representative and the caregiver
* Patients having participated in AFFiRiS 001 and received at least 1 vaccination with AFFITOPE AD01
* Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits.

Exclusion Criteria:

* Patients having received no vaccination with AFFITOPE AD01
* Contraindication for MRI imaging
* History of questionable compliance to visit schedule, patients not expected to complete the clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having participated in AFFiRiS 001, as AFFiRiS 003 is a follow-up trial.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Tolerability | 1 year

SECONDARY OUTCOMES:
Immunological and clinical efficacy (evaluated in an explorative manner only) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mueller, Univ. Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria